CLINICAL TRIAL: NCT00537173
Title: Predicting Response and Toxicity in Patients Receiving Paclitaxel and Avastin for Breast Cancer: A Multicenter Genomic, Proteomic and Pharmacogenomic Correlative Study
Brief Title: Predicting Response and Toxicity in Patients Receiving Paclitaxel and Avastin for Breast Cancer
Status: Terminated | Type: Observational
Why Stopped: Lack of Accrual
Sponsor: Hoosier Cancer Research Network (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Indiana University School of Medicine (Other); University of Colorado, Denver (Other); Baylor University (Other); McGill University (Other)
Responsible Party: Kathy Miller, M.D., Hoosier Oncology Group
Other Study IDs: HOG COE-02; DoD Grant BC030400 (Other: DoD)
Record Dates: First submitted 2007-09-26; First posted 2007-09-28 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy, Needle; Blood Specimen Collection; Paclitaxel; Bevacizumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tumor samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Arm 1: Paclitaxel 90 mg/m2 IV D1, 8, and 15 + Avastin 10 mg/kg IV, day 1 and 15
  Interventions: Procedure: Core Biopsy; Procedure: Blood Collection; Drug: Paclitaxel; Drug: Avastin

INTERVENTIONS:
Procedure: Core Biopsy — biopsy
Procedure: Blood Collection — Blood/serum sample
Drug: Paclitaxel — Paclitaxel 90 mg/m2 IV, day 1, 8 and 15
Drug: Avastin — Avastin 10 mg/kg IV, day 1 and 15

SUMMARY:
This trial provides a unique opportunity in that it combines genomic, proteomic and pharmacogenomic assessments in patients receiving chemotherapy for advanced breast cancer. To date no other trials have analyzed gene and protein expression at the same time points in the same patient, combined with clinical outcome. Similar to previous attempts to predict response based on expression of a single gene or protein, we expect that neither genomic or proteomic profiling alone will be sufficient to optimize therapy. Rather, we expect an iterative process that combines information gleaned from both platforms, modified to avoid toxicity based on pharmacogenomics.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

Sample Collection:

* Core biopsy
* Blood sample

  28-day Cycle Treatment Regimen:
* Paclitaxel 90 mg/m2 IV D1, 8, and 15
* Avastin 10 mg/kg IV D1 and 15

ECOG Performance Status of 0 or 1

Life Expectancy: Not specified

Hematopoietic:

* Platelet count > 100,000/mm³
* Absolute neutrophil count > 1200/mm³
* PTT < 1.5 x upper limit of normal
* INR < 1.5 x upper limit of normal

Hepatic:

* Total bilirubin < 1.5 mg/dL
* SGOT (AST) < 2 x upper limit of normal

Renal: Not specified

Cardiovascular:

* Clinically significant cardiovascular or cerebrovascular disease including prior myocardial infarction (within 6 months prior to study entry), unstable angina, Grade II or greater peripheral vascular disease, New York Heart Association (NYHA) Grade II or greater congestive heart failure, hypertensive crises, hypertensive encephalopathy or uncontrolled hypertension (SBP>150, DBP>100).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the breast with measurable locally recurrent, locally advanced (that is not amenable to resection with curative intent), or metastatic disease.
* Patients must consent to have a biopsy performed to obtain fresh tissue or be able to identify a FFPE tissue block in which tissue samples can be obtained to complete the testing for this study.
* Planned chemotherapy regimen of paclitaxel and Avastin for the treatment of metastatic breast cancer.
* Females age > 18 years
* Written informed consent and HIPAA authorization for release of personal health information.

Exclusion Criteria:

* Patients must not have had chemotherapy for locally recurrent or metastatic breast cancer.
* Hormonal therapy for locally recurrent or metastatic disease must have been discontinued at least 2 weeks prior to study entry.
* Patients must not have had adjuvant or neoadjuvant taxane therapy within 12 months prior to study entry.
* Breast cancer overexpressing HER-2 (gene amplification by FISH or 3+ overexpression by immunohistochemistry) are not eligible unless they have received prior therapy with Herceptin.
* Patients must not have had a major surgical procedure within 4 weeks prior to study entry. (Placement of vascular access device, and breast biopsy, will not be considered major surgery.)
* Patients must not have had a minor surgical procedure, placement of an access device, or fine needle aspiration within 7 days of starting protocol therapy.
* Patients must not have had radiation within 2 weeks prior to study entry.
* Previously radiated area(s) must not be the only site of disease for study entry.
* Patients must not have a history of bleeding diathesis or have used anticoagulant therapy within 10 days of study entry. (Low dose anticoagulant therapy to maintain patency of a vascular access device is allowed.)
* Patients with a history of deep vein thrombosis or pulmonary embolism are not eligible.
* Aspirin usage (> 325 mg/day) or other nonsteroidal anti-inflammatory medications known to inhibit platelet function daily are not allowed within 10 days prior to study entry.
* Patients currently using any of the following drugs known to inhibit platelet function are not eligible: dipyridamole (Persantine), ticlopidine (Ticlid), clopidogrel (Plavix) and cilostazol (Pletal).
* Patients must not have a history of TIA or CVA within 6 months prior to study entry.
* Patients must not have a history or radiologic evidence of CNS metastases including previously treated, resected or asymptomatic brain lesions or leptomeningeal involvement (head CT or MRI must be obtained within 6 weeks prior to study entry).
* Patients must not have a non-healing wound or fracture.
* Patients must not have a hypersensitivity to paclitaxel or drugs using the vehicle Cremophor, Chinese hamster ovary cell products or other recombinant human antibodies.
* Females must not be pregnant or breastfeeding. Females of childbearing potential must use an accepted and effective method of contraception (hormonal or barrier method of birth control; abstinence) while on treatment and for a 3 month period thereafter.
* Females of childbearing potential must have a negative pregnancy test within 7 days prior to being registered for protocol therapy. Subjects are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study entry
* Urine protein: creatinine (UPC) ratio > 1.0 at baseline or urine protein dipstick > 2+.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population is limited to patients with advanced breast cancer who are receiving paclitaxel + Avastin
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2007-09; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
To correlate tumor gene expression (genomic profile) with response to paclitaxel + Avastin in patients with advanced breast cancer | 36 months

SECONDARY OUTCOMES:
To correlate serum and tumor proteomic profiles with response; To compare serum and tissue proteomic analyses; To compare genomic and proteomic profiles; To correlate toxicity and/or response with drug-specific pharmacogenomic parameters. | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: George Sledge, M.D., Principal Investigator — Hoosier Oncology Group, Inc.
Locations (4):
- United States (4):
  - Cancer Care Center of Southern Indiana, Bloomington, Indiana
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Horizon Oncology Center, Lafayette, Indiana
  - Baylor College of Medicine - Methodist Breast Center, Houston, Texas

REFERENCES:
- See also: Hoosier Oncology Group Home Page — http://www.hoosieroncologygroup.org